CLINICAL TRIAL: NCT00354822
Title: Phase II Study for Use of Oral Fludarabine Plus Cyclophosphamide and Rituximab Followed by Zevalin as Front-Line Treatment for Non-Follicular Indolent Lymphomas.
Brief Title: Fludarabine,Cyclophosphamide and Rituximab Followed by Zevalin for Non-Follicular Indolent Lymphomas.
Acronym: Z0105
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit in time a sufficient number of patients
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Regional Hospital of Bolzano (Other)
Responsible Party: Corrado Tarella, MD, Gruppo Per Le Terapie Innovatove nei Linfomi (GITIL)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2005-000699-41
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Zevalin; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zevalin — Yttrium-90 (90Y) ibritumomab tiuxetan 0.4 mCi/kg is delivered to patient achieving at least a partial remission (PR) after chemotherapy as a single dose for patients with baseline platelet counts>150x10^9/L or 0.3 mCi/kg for patients with baseline platelet counts of 100 to 149x10^9/L. Rituximab 250mg/sqm is given prior to therapeutic radiolabeled antibodies.

SUMMARY:
Pilot multicentre, open label study with the aim to evaluate antitumor activity in term of the sum of complete and partial response (O.R.R.) of chemotherapy (cyclophosphamide and fludarabine) and rituximab, followed by zevalin radioimmunotherapy and response duration (Time to relapse or progression)and to evaluate the safety of the treatment as acute and late toxicity.

Secondary objective is to evaluate the overall survival (OS) and the event-free survival (EFS).

DETAILED DESCRIPTION:
Test medication:

* Yttrium-90 (90Y) ibritumomab tiuxetan 0.4 mCi/kg is delivered to patient achieving at least a partial remission (PR) after chemotherapy as a single dose for patients with baseline platelet counts>150x10^9/L or 0.3 mCi/kg for patients with baseline platelet counts of 100 to 149x10^9/L. Rituximab 250mg/sqm is given prior to therapeutic radiolabeled antibodies.
* Standard dose chemotherapy consisting of cyclophosphamide, fludarabine and rituximab given every 28 days up to the best response (maximum 6 courses).
* A prophylaxis for pneumocystis carinii as well as for herpes zoster are needed during treatment.

Main parameters of activity: activity of Yttrium-90 (90Y) ibritumomab tiuxetan after cyclophosphamide, fludarabine and rituximab combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a lymphoma refractory to front-line chemotherapy, not including fludarabine, or in first relapse after chemotherapy not including fludarabine, not suitable for high-dose chemotherapy supported by auto or allogeneic bone marrow transplantation.
* Histologically-confirmed small lymphocytic (SLL), lymphoplasmacytic (LPL) and marginal zone (MZL) lymphomas.
* All prior chemotherapy, including corticosteroids, had to have been completed > 4 weeks before study treatment; < 25% of active bone marrow irradiated previously; no prior bone marrow transplantation.
* Age: 18-70 years
* ECOG- performance status: 0-2.
* No allergy to mouse proteins.
* CD20 positive B cell lymphoma.
* Ann Arbor stage III or IV disease with bidimensionally measurable disease in at least one site which has not irradiated, including any adenopathy or mass that could be measured during a physical examination or that was > 5 cm on a computed tomographic scan (CT). In the event of splenomegaly or hepatomegaly, extension 5 cm below the costal margin was considered evidence of measurable disease. Osteoblastic bone lesions, ascites and pleural effusion are not considered measurable disease.
* Tumor involvement in the marrow<25% before treatment with Zevalin.
* Acceptable hematologic status within one week prior study start: Hb>9g/dL, white blood count >3x10^9/L, absolute neutrophil count >1.5x10^9/L, platelets >100x10^9/L.
* Written informed consent prior to any study specific screening procedures, with the understanding that the patient has the right to withdraw from that study at any time, without prejudice.
* Patients willing and able to comply with the protocol for the duration of the study.
* Patients, if sexually active, must agree to be using effective contraception for the entire treatment period and for 1 year following treatment. Women, of child-bearing potential, must have a negative pregnancy test.

Exclusion Criteria:

* Histologies other than those included
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of cervix within the last 5 years.
* Major surgery, other than diagnostic surgery, within the last 4 weeks.
* Presence of malignant ascites or pleural effusions.
* Evidence of CNS involvement. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmias not well controlled with medication, or myocardial infarction within the last 6 months, NYHA class III or IV heart disease), abnormal liver function tests, not disease related, within 1 week prior to study start (serum bilirubin >2 mg/dL; ALAT >2.5 x upper normal limit; alkaline phosphatase >2.5xupper normal limit), abnormal renal function, not disease related (serum creatinine >2.0 mg/dL), active opportunistic infections.
* Serum positivity for HIV, HBsAg and HCV except for those with no sign of active viral replication, assessed by HCV-RNA and HBV-DNA. This latter group of patients can be enrolled in the study, but they will receive lamivudine prophylaxis and bimonthly evaluation of HbSAg, HbCAb and HBV-DNA will be provided.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
achievement and duration of complete or partial reduction of lymphnodes six weeks after the end of treatment with zevalin | 2 years

SECONDARY OUTCOMES:
overall and event free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cortelazzo Sergio, MD, Principal Investigator — Ospedale Centrale di Bolzano (Italy)
Locations (6):
- Italy (6):
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo, BG
  - U.O. Ematologia Ospedali Civili Brescia, Brescia, BS
  - Medicina Nucleare ed Oncologia Medica AOU Policlinico Universitario di Messina, Messina, ME
  - Istituto per la Ricerca e la Cura del Cancro IRCC, Candiolo, TO
  - SC Ematologia 2 ASO S. Giovanni Battista, Torino, TO
  - U.O. Ematologia Ospedale Cà Foncello, Treviso, TV

REFERENCES:
- [Result] Brandt L, Kimby E, Nygren P, Glimelius B; SBU-group. Swedish Council of Technology Assessment in Health Care. A systematic overview of chemotherapy effects in indolent non-Hodgkin's lymphoma. Acta Oncol. 2001;40(2-3):213-23. doi: 10.1080/02841860151116286. PMID 11441933
- [Result] Solal-Celigny P, Brice P, Brousse N, Caspard H, Bastion Y, Haioun C, Bosly A, Tilly H, Bordessoule D, Sebban C, Harousseau JL, Morel P, Dupas B, Plassart F, Vasile N, Fort N, Leporrier M. Phase II trial of fludarabine monophosphate as first-line treatment in patients with advanced follicular lymphoma: a multicenter study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 1996 Feb;14(2):514-9. doi: 10.1200/JCO.1996.14.2.514. PMID 8636765
- [Result] Santini G, Nati S, Spriano M, Gallamini A, Pierluigi D, Congiu AM, Truini M, Rubagotti A, Chisesi T, Vimercati R, Rossi E, Sertoli MR, Mattei D, Marino G, Gobbi M. Fludarabine in combination with cyclophosphamide or with cyclophosphamide plus mitoxantrone for relapsed or refractory low-grade non-Hodgkin's lymphoma. Haematologica. 2001 Mar;86(3):282-6. PMID 11255275
- [Result] Hiddemann W, Dreyling M, Unterhalt M. Rituximab plus chemotherapy in follicular and mantle cell lymphomas. Semin Oncol. 2003 Feb;30(1 Suppl 2):16-20. doi: 10.1053/sonc.2003.50024. PMID 12652460
- [Result] Witzig TE, Flinn IW, Gordon LI, Emmanouilides C, Czuczman MS, Saleh MN, Cripe L, Wiseman G, Olejnik T, Multani PS, White CA. Treatment with ibritumomab tiuxetan radioimmunotherapy in patients with rituximab-refractory follicular non-Hodgkin's lymphoma. J Clin Oncol. 2002 Aug 1;20(15):3262-9. doi: 10.1200/JCO.2002.11.017. PMID 12149300
- [Result] Witzig TE, Gordon LI, Cabanillas F, Czuczman MS, Emmanouilides C, Joyce R, Pohlman BL, Bartlett NL, Wiseman GA, Padre N, Grillo-Lopez AJ, Multani P, White CA. Randomized controlled trial of yttrium-90-labeled ibritumomab tiuxetan radioimmunotherapy versus rituximab immunotherapy for patients with relapsed or refractory low-grade, follicular, or transformed B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2002 May 15;20(10):2453-63. doi: 10.1200/JCO.2002.11.076. PMID 12011122